CLINICAL TRIAL: NCT04783376
Title: Effect of Splitting Mealtime Insulin Doses Used for Mixed Meals High in Fat and Protein on Postprandial Blood Glucose Levels in Children and Adolescents With Type 1 Diabetes Mellitus Using Multiple Daily Injection Regimen
Brief Title: Effect of Splitting Mealtime Insulin Doses After Mixed Meals High in Fat and Protein
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sawsana Ewieda, Specialist registrar at Pediatrics Department, Sohag University Hospital, Sohag University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-01-02
Record Dates: First submitted 2021-02-24; First posted 2021-03-05 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (usual treatment) (Active Comparator): intervention A
  Interventions: Drug: : Insulin, lispro and regular insulin
- Arm 2(splitted bolus dose, fast-acting insulin only) (Active Comparator): intervention B
  Interventions: Drug: : Insulin, lispro and regular insulin
- Arm 3 (splitted bolus dose, fast acting insulin before the meal and regular insulin after the meal) (Active Comparator): intervention C
  Interventions: Drug: : Insulin, lispro and regular insulin

INTERVENTIONS:
Drug: : Insulin, lispro and regular insulin — * A: the participant will have a mealtime bolus dose of fast-acting insulin 10 minutes before the meal representing 100% of the dose calculated according to the carbohydrate content of the meal and the individual insulin to carbohydrate ratio
  * B: the bolus insulin dose for the meal will be calculated according to the carbohydrate content of the meal and the individual insulin to carbohydrate ratio and additional 30% of the calculated dose will added to cover the fat and protein content of the meal. This total dose will be divided into 2 portions. A premeal portion (60%) will be given 10 minutes before the meal and (40%) will be given 30 minutes after the premeal dose. Both doses will be given as fast-acting insulin.
  * C: the same as intervention B but the 40% of the total dose will be given as regular insulin.

SUMMARY:
The current management of type 1 diabetes mellitus (T1DM) depends on the use of intensive insulin therapy - either by insulin pump therapy or multiple daily injection (MDI) therapy - and the use of carbohydrate counting to determine the mealtime bolus insulin dose according the carbohydrate contents of each meal or snack. However, several studies reported that the fat and protein contents of the meals can also affect the postprandial blood glucose levels and result in delayed postprandial hyperglycemia especially after high fat and protein meals.

There is no widely accepted regimen to calculate insulin required for the fat and protein contents of meals especially for patients using multiple daily injection regimen. This study aims to find a better method to cover the increased insulin requirements following mixed fat and protein meals. The study will compare the effect of splitting mealtime bolus insulin doses into pre-meal and post-meal portions to the standard regimen which involve giving bolus dose depending on carbohydrate content only with additional correction doses 2 to 3 hours after the meal to compensate for the postprandial hyperglycemia induced by fat and protein content of the meals.

DETAILED DESCRIPTION:
The study will include children and adolescents aged 6 - 18 years, diagnosed with T1DM for at least 1 year, using multiple daily injection regimen and carbohydrate counting. The study participants will be admitted at the pediatric department, Sohag University Hospital for 1 week to adjust insulin doses. adjustments will be made to basal doses, insulin to carbohydrate ratio (ICR), insulin sensitivity factor (ISF) if required.

The study participants will have three test lunch meals on 3 consecutive days consumed at the pediatric department, Sohag university hospital at 12 PM. The test meals will consist of two slices of a deep pan pizza base topped with tomato sauce, mozzarella full fat soft cheese, and minced beef. (weight: 150 g, carb. 40 g, fat: 15 g, protein: 20 g, total calories 360 kcal). The meal will be consumed within 20 minutes.

Blood glucose level before the meal should be between 80 to 150 mg/dl. Correction doses can be given 3 hours before the test if needed to bring the blood glucose level to the desired target range before the test meals.

The participant will be assigned to use each one of the following interventions on a separate day in a random sequence.

* Intervention A: the participant will have a mealtime bolus dose of fast-acting insulin 10 minutes before the meal representing 100% of the dose calculated according to the carbohydrate content of the meal and the individual insulin to carbohydrate ratio (ICR). If hyperglycemia (blood glucose level >180 mg/dl) developed after 3 hours, the participant will receive an additional correction dose of fast-acting insulin calculated according to the individual insulin sensitivity factor (ISF).
* Intervention B: the bolus insulin dose for the meal will be calculated according to the carbohydrate content of the meal and the individual insulin to carbohydrate ratio (ICR) and additional 30% of the calculated dose will added to cover the fat and protein content of the meal. This total dose will be divided into 2 portions. A premeal portion (60% of the total dose) will be given 10 minutes before the meal. The remaining 40% of the total dose will be given 30 minutes after the premeal dose. Both doses will be given as fast-acting insulin.
* Intervention C: the bolus insulin dose for the meal will be calculated according to the carbohydrate content of the meal and the individual insulin to carbohydrate ratio (ICR) and additional 30% of the calculated dose will added to cover the fat and protein content of the meal. This total dose will be divided into 2 portions. A premeal portion (60% of the total dose) will be given 10 minutes before the meal as fast-acting insulin. The remaining 40% of the total dose will be given 30 minutes after the premeal dose as regular insulin.

Types of insulin: insulin lispro (Humalog 100 IU/mL) as fast-acting insulin and regular insulin (Humulin R) as regular insulin (Eli Lilly and Company, Indianapolis, IN, USA). Insulin doses will be calculated, splitted, approximated to the nearest 0.5 unit and given using Humapen Luxura half- unit increments insulin pens.

Capillary blood glucose level will be measured by a calibrated finger-prick blood glucose meter before the meals and every hour for the next 6 hours after the test meals. Moreover, venous blood glucose and serum cholesterol and triglycerides levels will be measured 3 hours after the test meals.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 6 - 18 years
* diagnosed with T1DM for at least 1 year
* using MDI regimen with advanced carbohydrate counting for at least 6 months

Exclusion Criteria:

* Subjects with associated

  * diabetic autonomic neuropathy
  * hypothyroidism
  * celiac disease.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose levels before the test meals. | before the test meals.
  Capillary blood glucose levels measured by a calibrated finger-prick blood glucose meter before the test meals
Capillary blood glucose levels one hour after the test meals. | one hour after the test meal
  Capillary blood glucose levels measured by a calibrated finger-prick blood glucose meter one hour after the test meals
Capillary blood glucose levels two hours after the test meals. | two hours after the test meal
  Capillary blood glucose levels measured by a calibrated finger-prick blood glucose meter two hours after the test meals
Capillary blood glucose levels three hours after the test meals. | three hours after the test meal
  Capillary blood glucose levels measured by a calibrated finger-prick blood glucose meter three hours after the test meals
Capillary blood glucose levels four hours after the test meals. | four hours after the test meal
  Capillary blood glucose levels measured by a calibrated finger-prick blood glucose meter four hours after the test meals
Capillary blood glucose levels five hours after the test meals. | five hours after the test meal
  Capillary blood glucose levels measured by a calibrated finger-prick blood glucose meter five hours after the test meals
Capillary blood glucose levels six hours after the test meals. | six hours after the test meal
  Capillary blood glucose levels measured by a calibrated finger-prick blood glucose meter six hours after the test meals

SECONDARY OUTCOMES:
assessment of serum cholesterol level three hours after the test meal following each intervention | 3 hours after test meal
  serum cholesterol levels measured 3 hours after the test meals.
assessment of serum triglyceride level three hours after the test meal following each intervention | 3 hours after test meal
  serum triglycerides levels measured 3 hours after the test meals.

CONTACTS AND LOCATIONS:
Locations (1):
- Sawsana Ewieda, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hegab AM, Hasaballah SE, Mohamed MM. Splitting Mealtime Insulin Doses for Mixed Fat and Protein Meals in Children and Adolescents with Type 1 Diabetes Using Multiple Daily Injection Regimen: A Randomized Cross-Over Trial. Pediatr Diabetes. 2023 Oct 27;2023:7467652. doi: 10.1155/2023/7467652. eCollection 2023. PMID 40303273